CLINICAL TRIAL: NCT01138644
Title: The "AFFORD" Study: Atrial Fibrillation/Flutter Outcome Risk Determination
Brief Title: Atrial Fibrillation/Flutter Outcome Risk Determination
Acronym: AFFORD
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Tyler Barrett, Assistant Professor of Emergency Medicine MD, MSCI, Vanderbilt University
Other Study IDs: The "AFFORD" Study; NHLBI (Other Grant/Funding Number: 1K23HL102069-01)
Record Dates: First submitted 2010-05-28; First posted 2010-06-07 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Atrial Fibrillation; Atrial Flutter
Keywords: Atrial Fibrillation; Atrial Flutter
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood for storing and conducting genetic testing.
Oversight: Data Monitoring Committee: No

SUMMARY:
It is our hypotheses that 1) readily available Emergency Department data can be utilized in an Atrial Fibrillation clinical prediction rule to identify those patients at low or high risk for adverse outcomes; 2) Assigned risk can be utilized to drive physician decision-making by identifying patients who do not require hospital admission (low risk) and patients needing hospitalization (high risk); and 3) a facile version of the AFPR will be easily incorporated into standard Emergency Department patient management systems and assist physicians with risk stratification of patients presenting with Atrial Fibrillation.

DETAILED DESCRIPTION:
AF: Impact on Present and Future National Health Over 2 million people in the United States have Atrial Fibrillation, the most common sustained arrhythmia.1 That number of patients is expected to increase to 5.6 million by 2050.1 Atrial Fibrillation is associated with a 4-5 fold increase in the risk of stroke, 3-fold increase in the risk of heart failure and 1.5-1.9 increased risk of death.2-6 The prevalence of Atrial Fibrillation increases as individuals age; 5.9% of those over 65 years of age and 9% of those over 80 years are diagnosed with the arrhythmia.25 The lifetime risk for development of Atrial Fibrillation is estimated to be 1 in 4 for men and women forty years of age and older.26 The proper management of patients with AF is critical due to the well-documented association with heart failure and stroke.2-6, 11, 27.

The number of Emergency Department visits for complaints related to Atrial Fibrillation increased by 88% between 1993 and 2003 and now account for approximately 1% percent of all Emergency Department visits in the United States.7, 24 More than 65% of these Atrial Fibrillation visits result in hospital admission and over $6.65 billion in expenditures, including $3.88 billion for hospitalizations, $1.53 billion for outpatient treatment and nearly $240 million for prescription drugs.8, 24 Patients with a primary admission diagnosis of AF had a mean length of stay and hospital charge of 4 days and $7000 in 1999.28 Over the past 20 years, the admission rate for Atrial Fibrillation has increased by 66%.29-31 The combination of increasing Atrial Fibrillation prevalence, unnecessarily high admission rate and Emergency Department crowding is likely to severely burden our healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* ED patients 18 years and older
* Provide informed consent
* Have a documented diagnosis of AF or atrial flutter on electrocardiogram or rhythm strip from an ED, prehospital provider or outside medical facility on day of enrollment.
* Present with signs (tachycardia, dyspnea) or symptoms (palpitations, chest pain, shortness of breath, weakness, lightheadedness, pre-syncope, or syncope) consistent with primary symptomatic AF
* Patients whose primary complaint is not directly related to their AF diagnosis (e.g. evaluation for febrile illness, gastrointestinal complaint, injury) BUT have a secondary complaint consistent with symptomatic AF that requires ED evaluation (e.g. new AF diagnosis, AF associated with inadequate rate control (defined as resting heart rate greater than 100bon), AF associated with heart failure symptoms, AF in the setting of CVA or TIA, AF associated with other thromboembolic complications).

Exclusion Criteria:

* Patients who are under the age of 18
* Previously enrolled patients
* ED patients who present with complaints unrelated to their AF (e.g. sprained ankle,pharyngitis) and have adequately rate (<100 bpm at rest) or rhythm controlled-AF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants for this study will be those with AF who present to the ED for their care. This study population will come from all walks of life and will not exclude any one group, sex, ethnicity, etc.
Sampling Method: Non-Probability Sample
Enrollment: 519 (Actual)
Dates: Start 2010-06; Primary Completion 2013-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Incidence of an atrial-fibrillation or atrial flutter related adverse event at 5 days from the index ED visit. | 5 days from ED visit
  We define adverse events as the following patient death, 5-day ED return visits and unscheduled hospital admissions for AF-related complaints, AF-related cardiovascular and thromboembolic complications.
Incidence of an Atrial fibrillation or atrial flutter related adverse event within 30 days of index ED visit | 30 days from ED visit
  We define adverse events as the following patient death, 30-day ED return visits and unscheduled hospital admissions for AF-related complaints, AF-related cardiovascular and thromboembolic complications.

SECONDARY OUTCOMES:
Patient death from any causes | 30 days
  We will record patient deaths due to any cause within 30 days of their ED visit. Only deaths classified as having cardiovascular causes will be included in the development of the prediction rule.

CONTACTS AND LOCATIONS:
Overall Officials: Tyler W Barrett, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center - Emergency Medicine, Nashville, Tennessee, United States

REFERENCES:
- [Background] Barrett TW, Storrow AB, Jenkins CA, Harrell FE Jr, Miller KF, Moser KM, Russ S, Roden DM, Darbar D. Atrial fibrillation and flutter outcomes and risk determination (AFFORD): design and rationale. J Cardiol. 2011 Sep;58(2):124-30. doi: 10.1016/j.jjcc.2011.06.007. Epub 2011 Aug 4. PMID 21820279
- [Result] Barrett TW, Storrow AB, Jenkins CA, Abraham RL, Liu D, Miller KF, Moser KM, Russ S, Roden DM, Harrell FE Jr, Darbar D. The AFFORD clinical decision aid to identify emergency department patients with atrial fibrillation at low risk for 30-day adverse events. Am J Cardiol. 2015 Mar 15;115(6):763-70. doi: 10.1016/j.amjcard.2014.12.036. Epub 2015 Jan 6. PMID 25633190
- [Result] Barrett TW, Jenkins CA, Self WH. Validation of the Risk Estimator Decision Aid for Atrial Fibrillation (RED-AF) for predicting 30-day adverse events in emergency department patients with atrial fibrillation. Ann Emerg Med. 2015 Jan;65(1):13-21.e3. doi: 10.1016/j.annemergmed.2014.08.023. Epub 2014 Sep 20. PMID 25245277
- [Derived] Barrett TW, Self WH, Darbar D, Jenkins CA, Wasserman BS, Kassim NA, Casner M, Shoemaker MB. Association of atrial fibrillation risk alleles and response to acute rate control therapy. Am J Emerg Med. 2016 Apr;34(4):735-40. doi: 10.1016/j.ajem.2016.01.034. Epub 2016 Feb 10. PMID 26920668